CLINICAL TRIAL: NCT04611321
Title: A Phase Ib/II, Open-Label, Single Arm Study to Evaluate the Safety and Efficacy of IBI318 in Participants With Advanced Cutaneous Squamous Cell Carcinoma.
Brief Title: Study of IBI318 in Patients With Advanced Cutaneous Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment, Innovent Biologics has decided not to continue this study after consultation with investigators.
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI318A201
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Advanced Cutaneous Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ib/II (Experimental): Patients with advanced CSCC. IBI318 administered intravenously every 2 weeks.
  Interventions: Drug: IBI318

INTERVENTIONS:
Drug: IBI318 — IBI318 will be given fixed dose via intravenous (IV) infusion on Day 1 of each 14-day cycle until disease progression or loss of clinical benefit.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of IBI318 (anti-PD-1/PD-L1) in adult participants with metastatic (nodal or distant) cutaneous squamous cell carcinoma (CSCC), or unresectable locally advanced CSCC that is not amenable to surgery and/or radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF.
2. Adults 18 years of age or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy at least 12 weeks.
5. Adequate organ and bone marrow function.
6. Histologically confirmed diagnosis of invasive CSCC. .

Exclusion Criteria:

1. Prior treatment with an agent that blocks the PD-1/PD-L1 pathway.
2. Any investigational drugs received within 4 weeks prior to the first study treatment.
3. Receive the last dose of anti-tumor therapy within 4 weeks before the first dose of study therapy.
4. History of autoimmune disease , present active autoimmune disease or inflammatory diseases
5. Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate ( evaluated by the independent review committee according to RECIST V1.1; 0-100%). Higher scores mean a better outcome | 24 months
  RECIST version 1.1 will be used to determine ORR by IRRC

SECONDARY OUTCOMES:
Investigator Assessments of Overall Response Rate | 24 months
  RECIST version 1.1 will be used to determine ORR by investigator
Duration of response | 24 months
  RECIST version 1.1 will be used to determine DOR by investigator and IRRC
PFS (progression-free survival) | 24 months
  RECIST version 1.1 will be used to determine PFS by investigator and IRRC
Overall Survival | 24 months
AEs and SAEs | 30 months
  To evaluate the safety and tolerability of IBI318 [Adverse events (AEs), Serious Adverse Events (SAEs) ]

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China